CLINICAL TRIAL: NCT03099278
Title: Ezetimibe for Patients With Chronic Hepatitis D
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziauddin Hospital (Other)
Responsible Party: Principal Investigator, Zaigham Abbas, Professor, Ziauddin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00281116ZAGE
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Chronic Hepatitis D
Keywords: hepatitis D; Ezetimibe; HDV RNA
MeSH Terms: conditions — Hepatitis D, Chronic; Hepatitis D | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ezetimibe (Experimental)
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe — Ezetimibe 20 mg oral daily

SUMMARY:
Ezetimibe possesses pharmacophore features to inhibit NTCP, the receptor required for HBV and HDV hepatocyte entry that include two hydrophobes and one hydrogen bond acceptor. Therapy with Ezetimibe may lead to decline in hepatitis D virus levels. The aim of the study is to evaluate the utility of Ezetimibe in patients with chronic HDV infection

ELIGIBILITY:
Inclusion Criteria:

* Treatment experienced patients; non-responders of relapsers of pegylated interferon therapy
* Age 18 years or above
* Presence of anti-HDV in serum
* Presence of quantifiable HDV RNA in serum
* Elevated ALT > ULN

Exclusion Criteria:

* Decompensated liver disease
* Patients with ALT levels greater than 10 times ULN (400 U/L)
* Pregnancy or inability to practice adequate contraception.
* Significant systemic or major illnesses other than liver disease, including, but not limited to, congestive heart failure, renal failure (eGFR<50 ml/min), organ transplantation, serious psychiatric disease or depression and active coronary artery disease.
* Systemic immunosuppressive therapy
* Evidence of another form of liver disease in addition to viral hepatitis
* Active substance abuse, such as alcohol or injection drugs
* Hepatocellular carcinoma
* Concurrent hepatitis C infection or HIV coinfection
* Diagnosis of malignancy in the five years
* Concurrent usage of statins
* Concurrent use of any other drug known to inhibit NTCP
* Inability to understand or sign informed consent
* Any other condition, which in the opinion of the investigators would impede the patient's participation or compliance in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
• Decline of HDV RNA quantitative measurements of >1 logs from baseline | 12 weeks of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Ziauddin University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No